CLINICAL TRIAL: NCT06496776
Title: The Effect of a Horizontal Apical Mattress Suturing Technique on the Width and Thickness of the Keratinized Mucosa After Dental Implant Surgery: A Clinical Trial
Brief Title: The Effect of a Suturing Technique on the Gingival Tissues Around Dental Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Collaborators: Al-Wataniya University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UDDS-OMFS-2-2024
Record Dates: First submitted 2024-07-04; First posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Edentulous Jaw; Missing Teeth; Gingival Diseases
MeSH Terms: conditions — Jaw, Edentulous; Anodontia; Gingival Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Choukroun's method (Experimental): Patients in this group will have a specific suturing technique (called Choukroun's method) after dental implant insertion.
  Interventions: Procedure: Choukroun's technique

INTERVENTIONS:
Procedure: Choukroun's technique — Suturing will be done using the method described by Choukroun.

SUMMARY:
There is general agreement that a thick zone of the keratinized tissues around implants promotes accurate prosthetic procedures, permits oral hygiene maintenance, resists recession, and enables esthetic blending with surrounding tissues. A new procedure called Choukroun's technique has been suggested, and it consists of a combination of horizontal apical mattress suture with regular suture to increase the keratinized tissue in the mandibular arch during the first stage after implantation. The proposed procedure has not been evaluated yet in a cohort of patients. Therefore, this study aimed to evaluate the impact of Choukroun's technique on the width and thickness of the keratinized gingiva after oral surgery.

DETAILED DESCRIPTION:
A clinical trial will be conducted on patients referred to the Department of Oral and Maxillofacial Surgery at the Faculty of Dentistry, Al-Wataniya Private University, who have been referred to undergo dental implant surgery. The inclusion criteria for the study group were as follows: patients with mandibular missing teeth, good oral health, good general health, 18 to 70 years old, at least 1 mm thickness of keratinized gingiva, and at least 1 mm width of the attached gingiva. A total of 14 patients aged 27 to 67 years will be included in the study. After inserting the dental implants, the suturing will be conducted according to Choukroun's method.

The width and thickness of the keratinized gingiva will be assessed before surgery and at one and two months post-surgery. Repeated measures Analysis of Variance (ANOVA) will be applied to detect significant differences between assessment times.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mandibular missing teeth
* Good oral health
* Good general health
* Male or female
* Age between 18 and 70 years old,
* Thickness of the keratinized gingiva is at least 1 mm,
* The width of the attached gingiva is at least 1 mm.

Exclusion Criteria:

* Patients who are smokers
* Pregnant or lactating women
* Patients with systemic diseases
* Patients who have been taking medication in the last six months that could influence wound healing after surgery and
* Patients with oral inflammation such as periodontal disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-02-13 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
Change in the width of the keratinized gingiva | This variable will be measured at one day before surgery (T0), at one month (T1) and two months (T2) after the implant surgical insertion.
  The width of the attached gingiva will be measured using a periodontal probe (William's probe). This measurement will be made at the mesial, distal, and middle positions within the surgical area (from the crest of the alveolar ridge to the mucogingival junction), and the mean of these measurements will be recorded.
Change in the thickness of the keratinized gingiva | This variable will be measured at one day before surgery (T0), at one month (T1) and two months (T2) after the implant surgical insertion.
  To measure the thickness of the keratinized gingiva, an endodontic file equipped with a rubber tip will be used to penetrate the gingiva at various points within the surgical area until it reaches the bone surface. These points are located midway between the mid-crestal of keratinized gingiva and the mucogingival junction, spaced 2 millimeters apart, and extending from the mesial to the distal aspects of the surgical area. The thickness will be then measured using a ruler, and the mean of these values will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Khaled Abou-Agwa, DDS MSc PhD, Principal Investigator — Department of Oral and Maxillofacial Surgery, College of Dentistry, Al-Wataniya Private University
Locations (1):
- Department of Oral and Maxillofacial Surgery, Hama, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Silverstein LH, Kurtzman GM, Shatz PC. Suturing for optimal soft-tissue management. J Oral Implantol. 2009;35(2):82-90. doi: 10.1563/1548-1336-35.2.82. PMID 19400063
- [Background] Banche G, Roana J, Mandras N, Amasio M, Gallesio C, Allizond V, Angeretti A, Tullio V, Cuffini AM. Microbial adherence on various intraoral suture materials in patients undergoing dental surgery. J Oral Maxillofac Surg. 2007 Aug;65(8):1503-7. doi: 10.1016/j.joms.2006.10.066. PMID 17656275
- [Background] Rodeheaver GT, Beltran KA, Green CW, Faulkner BC, Stiles BM, Stanimir GW, Traeland H, Fried GM, Brown HC, Edlich RF. Biomechanical and clinical performance of a new synthetic monofilament absorbable suture. J Long Term Eff Med Implants. 1996;6(3-4):181-98. PMID 10167360
- [Background] Lee WH, Kuchler U, Cha JK, Stavropoulos A, Lee JS. Distance of insertion points in a mattress suture from the wound margin for ideal primary closure in alveolar mucosa: an in vitro experimental study. J Periodontal Implant Sci. 2021 Jun;51(3):189-198. doi: 10.5051/jpis.2100680034. PMID 34114382